CLINICAL TRIAL: NCT06408207
Title: Randomized Control Trial Evaluating the Impact of CGM Academy Education Curriculum Versus Standard Care on Glycemic Outcomes for Youth With Type 1 Diabetes
Brief Title: CGM Academy for Youth With Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Barber, Rebecca, Principal Investigator, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-23-00298
Record Dates: First submitted 2023-05-22; First posted 2024-05-10 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-07

CONDITIONS: Type1 Diabetes
Keywords: Continuous Glucose Monitoring; Glycemic Control; Diabetes Education; Type1 Diabetes

STUDY DESIGN:
Intervention Model Description: Simple randomization
Masking Description: Everyone will know their assigned intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CGM Academy (Experimental): * receive an interactive workbook with problem-based learning scenarios and video links about CGM and glucose management strategies.
  * participate in four in-depth online group sessions with diabetes care and education specialists
  * complete questionnaires three times: at the time of study enrollment, week 4 and 6 months.
  Interventions: Behavioral: CGM Academy
- Standard Diabetes Education (No Intervention): * receive standard education provided to all patients at CHLA
  * complete questionnaires three times: at the time of study enrollment, week 4 and 6 months.

INTERVENTIONS:
Behavioral: CGM Academy — Educational materials as well as online sessions with diabetes educators.
  Arms: CGM Academy

SUMMARY:
The goal of this randomized clinical trial is to compare the effects of a virtual education curriculum in blood glucose variation of youth with type 1 diabetes wearing continuous glucose monitoring (CGM) device. The main questions the study aims to answer are:

* Do participants undertaking the proposed curriculum present improved glucose variation than participants of standard education?
* Explore relationships between participant's glycemic outcomes with diabetes distress, diabetes family responsibilities, and number of hours of diabetes education.

Participants in the intervention group will:

* receive an interactive workbook with problem-based learning scenarios and video links about CGM and glucose management strategies.
* participate in four in-depth online group sessions with diabetes care and education specialists
* complete questionnaires three times: at the time of study enrollment, week 4 and 6 months.

Participants in the comparison group will:

* receive standard education provided to all patients at CHLA
* complete questionnaires three times: at the time of study enrollment, week 4 and 6 months.

DETAILED DESCRIPTION:
Youth with type 1 diabetes (T1D) are at increased risk for kidney failure, vision loss, heart disease, and premature mortality due to challenges with glycemic excursions. Continuous glucose monitoring (CGM) systems represent an important advance in diabetes technology with significant advantages over self-monitored blood glucose and the potential to optimize glycemic management. Despite these advances, youth with T1D, including patients at Children's Hospital Los Angeles (CHLA), fail to achieve recommended glycemic targets, highlighting the opportunity for testing innovative diabetes education programs aimed at increased technology uptake such as the CGM Academy intervention.

ELIGIBILITY:
Inclusion Criteria:

* Current age of 8-18 years, age group eligible for CGM therapy with Dexcom G6 and G7
* T1D duration ≥6 months, as insulin adjustments during honeymoon stage differs from establishedT1D
* Able to speak, read, and write English or Spanish
* Smartphone compatible with Dexcom G6 and G7application
* Ability to participate in virtual visits

Exclusion Criteria:

• Known history of medical adhesive allergies

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean change in Hemoglobin A1c from baseline to 6 months | Baseline to 6 months
  Change in Hemoglobin A1c

SECONDARY OUTCOMES:
Mean change in HbA1c (%) from baseline to 6 months. | Baseline to 6 months
  Change in Hemoglobin A1c
Mean change in CGM metrics measured by CGM readings | Week 4 & 6 months
  % Glucose Time in Range (70-180 mg/dL), % Glucose Time Below Range (<70mg/dL), % Glucose Time Above Range (>180mg/dL).
Change in perceived diabetes distress at baseline, week 4 & 6 months | Baseline, Week 4 & 6 months
  The Problem Areas in Diabetes survey (PAID) is an 18-item survey to assess the perceived burden associated with diabetes. Youth and caregivers are given statements about diabetes-related issues and report on a 5-point Likert scale (0 = not a problem, 1 = minor problem, 2 = moderate problem, 3 = somewhat serious problem, 4 = serious problem) the degree to which the statements are a problem for them. Increasing scores denote increased burden perceived.
Change in perceived diabetes family responsibility at baseline, week 4 & 6 months. | Baseline, week 4 & 6 months
  The Diabetes Family Responsibility Questionnaire (DFRQ) is a 14-item validated survey assessing parental and child involvement in various diabetes management tasks. Youth and caregivers report on a 3-point scale (1=child, 2=equal, 3=parent) who is responsible for a given diabetes task. Higher scores indicate more parental involvement in diabetes management.
Average number of diabetes educator hours used per study participant at week 4 & 6 months. | Week 4 and 6 months
  Number of hours spent in diabetes education
Perceived benefits of Continuous Glucose Monitor (CGM) use | week 4 & 6 months
  Adolescent Benefits and Burdens of CGM Survey - BenCGM & BurCGM. Participants answer each question on a scale of Strong Disagree, Disagree, Neutral, Agree, Strongly Agree.
Perceived burden of Continuous Glucose Monitor (CGM) use | week 4 & 6 months
  Adolescent Benefits and Burdens of CGM Survey - BenCGM & BurCGM. Participants answer each question on a scale of Strong Disagree, Disagree, Neutral, Agree, Strongly Agree.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Barber, PhD, RN, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No